CLINICAL TRIAL: NCT02449889
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre Trial Comparing the Efficacy and Safety of Highly Purified Human Chorionic Gonadotropin (HP-hCG) and Recombinant Human Chorionic Gonadotropin (rhCG) for Triggering of Final Follicular Maturation in Women Undergoing Controlled Ovarian Stimulation
Brief Title: A Randomised Trial Using Highly Purified Human Chorionic Gonadotropin (HP-hCG) and Recombinant Human Chorionic Gonadotropin (rhCG) in Women Undergoing Controlled Ovarian Stimulation
Acronym: FASHION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000191
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HP-hCG IM (Experimental): highly purified human chorionic gonadotropin, intramuscularly (IM)
  Interventions: Drug: highly purified human chorionic gonadotropin
- HP-hCG SC (Experimental): highly purified human chorionic gonadotropin, subcutaneously (SC)
  Interventions: Drug: highly purified human chorionic gonadotropin
- rhCG (Active Comparator): recombinant human chorionic gonadotropin
  Interventions: Drug: recombinant human chorionic gonadotropin

INTERVENTIONS:
Drug: highly purified human chorionic gonadotropin
  Other Names: CHORAPUR; BREVACTID
  Arms: HP-hCG IM; HP-hCG SC
Drug: recombinant human chorionic gonadotropin
  Other Names: OVIDREL; OVITRELLE
  Arms: rhCG

SUMMARY:
This trial is investigating the efficacy and safety of highly purified human chorionic gonadotropin (HP-hCG) and recombinant human chorionic gonadotropin (rhCG) for triggering of final follicular maturation in women undergoing controlled ovarian stimulation

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females between the ages of 18 and 39 years
* Documented history of infertility
* Body mass index (BMI) between 17.5 and 32.0 kg/m2
* Regular menstrual cycles

Exclusion Criteria:

* Known endometriosis stage III and IV
* Known polycystic ovarian syndrome (PCOS)
* History of recurrent miscarriage
* History of more than three previous controlled ovarian stimulation cycles

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07-09 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Instituto Ideia Fértil de Saúde Reproductive (there may be other sites in this country), São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 sites in Brazil randomized subjects to the trial.
Pre-assignment Details: In total 245 subjects were screened. Of these, 69 were screening failures and 176 were randomized. All randomized subjects were exposed to investigational medicinal product (IMP).
Groups:
- HP-hCG IM: Highly purified human chorionic gonadotropin 5000 international units (IU), intramuscularly (IM)
  Highly purified human chorionic gonadotropin
- HP-hCG SC: Highly purified human chorionic gonadotropin, 5000 IU subcutaneously (SC)
  Highly purified human chorionic gonadotropin
- rhCG SC: Recombinant human chorionic gonadotropin 250 µg SC
  Recombinant human chorionic gonadotropin
Period: Overall Study
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Started | 58 | 58 | 60
Completed | 57 | 52 | 59
Not Completed | 1 | 6 | 1
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) analysis set was defined as all randomized subjects. Subjects were analyzed according to planned (randomized) treatment. All relevant baseline data were summarized based on the ITT analysis set. The ITT analysis set included all 176 randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC | Total
Number analyzed (Participants) | 58 | 58 | 60 | 176
Age, Customized [Count of Participants; unit: Participants]
  <35 years | 35 | 33 | 32 | 100
  35-37 years | 20 | 23 | 22 | 65
  >=38 years | 3 | 2 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 60 | 176
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 10 | 23
  White | 49 | 51 | 50 | 150
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 58 | 58 | 60 | 176

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: Oocyte retrieval took place 36 h (±2h) after hCG administration. At oocyte retrieval the number of oocytes retrieved was recorded.
Time Frame: Approximately 36 hours after hCG administration
Population: The ITT analysis set was defined as all randomized subjects. Subjects were analyzed according to planned (randomized) treatment.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
Number of oocytes | 7.1 (4.6) | 7.3 (4.8) | 6.6 (4.1)
Statistical Analysis 1: Comparison: HP-hCG IM vs rhCG SC; Mean number of oocytes retrieved for the treatment comparison of HP-hCG IM versus rhCG SC; Test type: Non-Inferiority — Treatment comparisons were done in a sequential manner. First non-inferiority (NI) was tested for HP-hCG IM compared to rhCG SC (lower limit of the 95% confidence interval (CI) > -3.0). If NI was demonstrated, NI was also to be tested for HP-hCG SC compared to rhCG SC; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.8] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors
Statistical Analysis 2: Comparison: HP-hCG SC vs rhCG SC; Mean number of oocytes retrieved for the treatment comparison of HP-hCG SC versus rhCG SC; Test type: Non-Inferiority — As step 2 in the pre-specified sequential testing, NI was tested for HP-hCG SC compared to rhCG SC; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.5 to 2.0] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors

2. Secondary Outcome: Number of Metaphase II (MII) Oocytes
Description: Only applicable for insemination using intracytoplasmic sperm injection (ICSI). The MII oocytes were counted prior to insemination.
Time Frame: Prior to insemination (within 6 hours after oocyte retrieval)
Population: The ITT analysis set was defined as all randomized subjects. Subjects were analyzed according to planned (randomized) treatment.
  Note that only subjects with ICSI were included in this analysis, i.e. 58 subjects in the HP-hCG IM group, 55 subjects in the HP-hCG SC group and 57 subjects in the rhCG SC group.
Measure: Mean (Standard Deviation); unit: Number of MII oocytes
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 55 | 57
Number of MII oocytes | 5.9 (3.7) | 6.2 (3.5) | 5.6 (3.3)
Statistical Analysis 1: Comparison: HP-hCG IM vs rhCG SC; Number of MII oocytes retrieved for the treatment comparison of HP-hCG IM versus rhCG SC; Test type: Non-Inferiority — Pre-specified supportive endpoint analyzed in a similar manner as the primary endpoint; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.6 to 1.5] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors
Statistical Analysis 2: Comparison: HP-hCG SC vs rhCG SC; Number of Mll oocytes retrieved for the treatment comparison of HP-hCG SC versus rhCG SC; Test type: Non-Inferiority — Pre-specified supportive endpoint analyzed in a similar manner as the primary endpoint; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.4 to 1.6] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors

3. Secondary Outcome: Number of Fertilized (2 Pronuclei (2PN)) Oocytes
Description: Fertilization was assessed by counting the number of pronuclei, which was recorded as 0, 1, 2 or >2. Correct fertilization was defined as oocytes with 2PN.
Time Frame: One day after oocyte retrieval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of fertilized oocytes
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
Number of fertilized oocytes | 4.4 (3.3) | 4.7 (3.4) | 4.2 (2.7)
Statistical Analysis 1: Comparison: HP-hCG IM vs rhCG SC; Number of fertilized (2 pronuclei (2PN)) oocytes for the treatment comparison of HP-hCG IM versus rhCG SC; Test type: Non-Inferiority — Pre-specified supportive endpoint analyzed in a similar manner as the primary endpoint; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.6 to 1.3] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors
Statistical Analysis 2: Comparison: HP-hCG SC vs rhCG SC; Number of fertilized (2 pronuclei (2PN)) oocytes for the treatment comparison of HP-hCG SC versus rhCG SC; Test type: Non-Inferiority — Pre-specified supportive endpoint analyzed in a similar manner as the primary endpoint; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.5 to 1.4] — ANOVA with treatment, stratum (<10 or ≥10 follicles with a diameter ≥12 mm), and site as fixed factors

4. Secondary Outcome: Positive β Unit of Human Chorionic Gonadotropin (βhCG) Rate
Description: Defined as percentage of subjects with positive beta hCG. A positive β hCG was confirmed by a blood test obtained 13-15 days after transfer.
Time Frame: 13-15 days after transfer
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
percentage of participants | 50.0 | 37.9 | 36.7

5. Secondary Outcome: Clinical Pregnancy Rate
Description: Defined as percentage of subjects with clinical pregnancy. Clinical pregnancy was defined as at least one gestational sac 5-6 weeks after transfer.
Time Frame: 5-6 weeks after transfer
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
percentage of participants | 46.6 | 27.6 | 31.7

6. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: The number of treatment-emergent AEs (TEAEs) in each treatment group will be presented.
Time Frame: AEs were collected from signing informed consent until end of trial visit = maximum period approximately 5 months. However, only TEAEs are presented
Population: Safety was summarized based on the safety analysis set.The safety analysis set included all 176 subjects. Subjects were analyzed according to their actual treatment.
Measure: Number; unit: Number of AEs
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
Number of AEs | 22 | 25 | 25

7. Secondary Outcome: Intensity of AEs
Description: The intensity of an TEAE would be classified using the following 3-point scale: mild (awareness of signs or symptoms, but no disruption of usual activity), moderate (event sufficient to affect usual activity [disturbing]) or severe (inability to work or perform usual activities [unacceptable]).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG SC
Number analyzed (Participants) | 58 | 58 | 60
Participants
  Any mild AE | 14 | 18 | 22
  Any moderate AE | 8 | 6 | 3
  Any severe AE | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from signing informed consent until end of trial visit = maximum period approximately 5 months.
Description: AEs with onset after IMP administration were considered treatment-emergent and are presented for the safety analysis set.
Groups:
- rhCG: Recombinant human chorionic gonadotropin 250 µg SC
  Recombinant human chorionic gonadotropin
Arm/Group | HP-hCG IM | HP-hCG SC | rhCG
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/58 | 2/60
Other Adverse Events (participants affected / at risk) | 12/58 | 12/58 | 11/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP-hCG IM (N=58) | HP-hCG SC (N=58) | rhCG (N=60)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP-hCG IM (N=58) | HP-hCG SC (N=58) | rhCG (N=60)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 6 (6) | 3 (3)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 3 (3)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 1 (2)
Vanishing twin syndrome (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator (PI) is that Sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the Sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Sponsor to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02449889/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT02449889/SAP_001.pdf